CLINICAL TRIAL: NCT05303324
Title: A Phase 1, Randomized, Open-Label, 2-Way Crossover Study to Assess the Single-Dose Pharmacokinetics of ALXN1840 Enteric-Coated Tablets at 2 Dose Strengths in Healthy Adult Subjects
Brief Title: Study of Oral ALXN1840 at 2 Dose Strengths in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN1840-HV-104; 2019-000516-28 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: ALXN1840; Enteric-coated tablet; Pharmacokinetics; Pharmacodynamics; Healthy
MeSH Terms: interventions — tetrathiomolybdate; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence 1 (AB) (Experimental): Participants received ALXN1840 once in each Period as a single oral dose under fasted conditions as follows:
  Period 1: ALXN1840 as a single EC tablet (Treatment A, reference). Period 2: ALXN1840 as three EC tablets (Treatment B, test).
  Participants were discharged following the 240-hour post-dose procedures (approximately 10 days after dosing in each period) unless it was medically necessary to extend the confinement.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840
- Sequence 2 (BA) (Experimental): Participants received ALXN1840 once in each Period as a single oral dose under fasted conditions as follows:
  Period 1: ALXN1840 as three EC tablets (Treatment B, test). Period 2: ALXN1840 as a single EC tablet (Treatment A, reference).
  Participants were discharged following the 240-hour post-dose procedures (approximately 10 days after dosing in each period) unless it was medically necessary to extend the confinement.
  There was a washout period of at least 14 days between each ALXN1840 dosing.
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — Participants received ALXN1840 at Hour 0 on Day 1 of the dosing period.
  Other Names: Bis-choline Tetrathiomolybdate; Tiomolibdic Acid; WTX101 (formerly)

SUMMARY:
To assess the relative bioavailability of ALXN1840 administered orally as a single enteric-coated (EC) tablet (reference, Treatment A) versus three EC tablets (test, Treatment B).

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≤ 100 kilograms (kg) and body mass index within the range 18-25 kg/meter squared, inclusive, at Screening.
* Negative serum pregnancy test at Screening and Day -1 for all women of childbearing potential.
* Willing to adhere to contraception requirements.
* Satisfactory medical assessment with no clinically significant or relevant abnormalities.

Exclusion Criteria:

* Current or recurrent/chronic disease
* Positive test for hepatitis B surface antigen or human immunodeficiency virus antibody at Screening.
* Acute or chronic hepatitis C virus infection.
* History of hypersensitivity to ALXN1840 or its excipients or any significant allergic reaction.
* Use of prescription medications (excluding oral contraceptives) within 14 days prior to dosing on Day 1, except with prior approval of the Sponsor.
* Participation (that is, last protocol-required study visit) in a clinical study within 90 days before initiation of dosing on Day 1.
* Serum ceruloplasmin value outside of the normal range at Screening
* Female participants who were breastfeeding.
* Prior exposure to ALXN1840.
* Major surgery or hospitalization within 90 days prior to dosing on Day 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 2 treatment sequences (A-B) or (B-A) in a crossover study design during 2 dosing periods. Participants were scheduled to receive either treatment A or B on Day 1 of each dosing period. There was a washout of at least 14 days between the dosing periods.
Groups:
- ALXN1840 Treatment Sequence A-B: Period 1: Participants received ALXN1840 reference formulation administered orally as 1 enteric-coated (EC) tablet at 15 milligrams (mg) on Day 1 (Treatment A).
  Period 2: Participants received ALXN1840 test formulation administered orally as 3 EC tablets at 5 mg (15 mg total) on Day 1 (Treatment B). There was a washout of at least 14 days between the dosing periods.
- ALXN1840 Treatment Sequence B-A: Period 1: Participants received ALXN1840 test formulation administered orally as 3 EC tablets at 5 mg (15 mg total) on Day 1 (Treatment B).
  Period 2: Participants received ALXN1840 reference formulation administered orally as 1 EC tablet at 15 mg on Day 1 (Treatment A). There was a washout of at least 14 days between the dosing periods.
Period: Treatment Period 1
Arm/Group | ALXN1840 Treatment Sequence A-B | ALXN1840 Treatment Sequence B-A
Started | 25 | 23
Received at Least 1 Dose of Study Drug | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | ALXN1840 Treatment Sequence A-B | ALXN1840 Treatment Sequence B-A
Started | 25 | 23
Received at Least 1 Dose of Study Drug | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- ALXN1840 Treatment Sequence A-B: Period 1: Participants received ALXN1840 reference formulation administered orally as 1 EC tablet at 15 mg on Day 1 (Treatment A).
  Period 2: Participants received ALXN1840 test formulation administered orally as 3 EC tablets at 5 mg (15 mg total) on Day 1 (Treatment B). There was a washout of at least 14 days between the dosing periods.
- Total: Total of all reporting groups
Arm/Group | ALXN1840 Treatment Sequence A-B | ALXN1840 Treatment Sequence B-A | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.63) | 28.1 (6.04) | 28.4 (6.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 0 | 2
  Race: Black or African American | 2 | 3 | 5
  Race: White | 18 | 18 | 36
  Race: Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed (Plasma) Concentration (Cmax) of Total Molybdenum
Description: The pharmacokinetic (PK) data of plasma total molybdenum were analyzed in the scope of this study as a surrogate measure for ALXN1840. Whole blood samples were collected for the measurement of plasma concentrations of total molybdenum via inductively coupled plasma-mass spectroscopy (ICP-MS).
Time Frame: Up to 240 hours postdose
Population: The Pharmacokinetic Population included all participants who had sufficient plasma samples to enable the calculation of PK parameters of at least the area under the plasma concentration versus time curve (AUC) for at least 1 Treatment Period. Participants were grouped by period for each treatment for this analysis.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Groups:
- ALXN1840 Treatment A: Participants received ALXN1840 reference formulation administered orally as 1 EC tablet at 15 mg on Day 1.
- ALXN1840 Treatment B: Participants received ALXN1840 test formulation administered orally as 3 EC tablets at 5 mg (15 mg total) on Day 1.
Arm/Group | ALXN1840 Treatment A | ALXN1840 Treatment B
Number analyzed (Participants) | 48 | 48
nanograms (ng)/milliliter (mL) | 173.10 (78.098) | 174.27 (62.956)

2. Primary Outcome: Area Under The Plasma Concentration Versus Time Curve From Time 0 (Dosing) to the Last Quantifiable Concentration (AUCt) of Total Molybdenum
Description: The PK data of plasma total molybdenum were analyzed in the scope of this study as a surrogate measure for ALXN1840. Whole blood samples were collected for the measurement of plasma concentrations of total molybdenum via ICP-MS.
Time Frame: Up to 240 hours postdose
Population: The Pharmacokinetic Population included all participants who had sufficient plasma samples to enable the calculation of PK parameters of at least the AUC for at least 1 Treatment Period. Participants were grouped by period for each treatment for this analysis.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | ALXN1840 Treatment A | ALXN1840 Treatment B
Number analyzed (Participants) | 48 | 48
hours*ng/mL | 7054.5 (3634.92) | 6990.5 (3020.70)

3. Secondary Outcome: Number of Participants With a Treatment-Emergent Adverse Event (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE was an AE that started during or after the first dose, or started prior to the first dose and increased in severity after the first dose. A related TEAE was defined as having a reasonable possibility the study intervention caused the AE as assessed by the investigator. Serious AEs (SAEs) were defined as any untoward medical occurrence that met at least 1 of the following serious criteria: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, other medically important serious event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 43
Population: The Safety Population included all participants who received at least 1 dose of study drug. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: ALXN1840 Treatment A; Period 2: ALXN1840 Treatment A: Participants received ALXN1840 reference formulation administered orally as 1 EC tablet at 15 mg on Day 1.
- Period 1: ALXN1840 Treatment B; Period 2: ALXN1840 Treatment B: Participants received ALXN1840 test formulation administered orally as 3 EC tablets at 5 mg (15 mg total) on Day 1.
Arm/Group | Period 1: ALXN1840 Treatment A | Period 1: ALXN1840 Treatment B | Period 2: ALXN1840 Treatment A | Period 2: ALXN1840 Treatment B
Number analyzed (Participants) | 25 | 23 | 23 | 25
Participants
  Any TEAE | 7 | 5 | 4 | 8
  Any serious TEAE (SAE) | 0 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 0 | 0
  Any related TEAE | 4 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 43
Description: The Safety Population included all participants who received at least 1 dose of study drug. Participants were analyzed as randomized.
Arm/Group | Period 1: ALXN1840 Treatment A | Period 1: ALXN1840 Treatment B | Period 2: ALXN1840 Treatment A | Period 2: ALXN1840 Treatment B
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 7/25 | 5/23 | 4/23 | 8/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: ALXN1840 Treatment A (N=25) | Period 1: ALXN1840 Treatment B (N=23) | Period 2: ALXN1840 Treatment A (N=23) | Period 2: ALXN1840 Treatment B (N=25)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05303324/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT05303324/SAP_001.pdf